CLINICAL TRIAL: NCT03525886
Title: A Phase 2, Open-Label, Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NBI-74788 in Adult Subjects With Congenital Adrenal Hyperplasia
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NBI-74788 in Adults With Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NBI-74788-CAH2001
Record Dates: First submitted 2018-05-02; First posted 2018-05-16 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: CAH - Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — crinecerfont

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (50 mg QHS) (Experimental): NBI-74788 50 mg once daily at bedtime (QHS) administered orally for 14 consecutive days.
  Interventions: Drug: NBI-74788
- Cohort 2 (100 mg QHS) (Experimental): NBI-74788 100 mg once daily at bedtime (QHS) administered orally for 14 consecutive days.
  Interventions: Drug: NBI-74788
- Cohort 3 (100 mg QPM) (Experimental): NBI-74788 100 mg once daily in the evening (QPM) administered orally for 14 consecutive days.
  Interventions: Drug: NBI-74788
- Cohort 4 (100 mg BID) (Experimental): NBI-74788 100 mg twice daily (BID) administered orally for 14 consecutive days.
  Interventions: Drug: NBI-74788

INTERVENTIONS:
Drug: NBI-74788 — Capsule, administered daily.

SUMMARY:
This is a Phase 2, open-label, multiple-dose, dose-escalation study to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of NBI-74788 in up to 30 adult female and male subjects (18 to 50 years of age) with a documented medical diagnosis of classic 21-hydroxylase deficiency congenital adrenal hyperplasia (CAH). The study will include a sequential-cohort design with four NBI-74788 dosing regimens, with each regimen administered for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Be in good general health.
2. Have a medically confirmed diagnosis of classic 21-hydroxylase deficiency CAH.
3. Be on a stable regimen of steroidal treatment for CAH that is expected to remain stable throughout the study.
4. Subjects of childbearing potential must be instructed on the proper use of barrier methods of contraception and agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently from screening until the final study visit or a prespecified window after the last dose of study drug, whichever is longer.
5. Subjects of childbearing potential must have a negative pregnancy test at screening and negative urine pregnancy test at baseline.
6. Have a negative urine drug (for illegal drugs) and alcohol breath test at screening and baseline.
7. Be willing and able to adhere to the study regimen and study procedures described in the protocol and informed consent/assent form, including all requirements at the study center and return for the follow-up visit.
8. Be willing to provide authorization for access to personal health information in conjunction with US Health Insurance Portability and Accountability Act (HIPAA).

Exclusion Criteria:

1. Have a clinically significant unstable medical condition or chronic disease, or malignancy.
2. Had a medically significant illness within 30 days of screening.
3. Have a known or suspected differential diagnosis of any of the other known forms of classic CAH.
4. Have a history that includes bilateral adrenalectomy, hypopituitarism, or other condition requiring daily therapy with orally administered glucocorticoids.
5. Are pregnant or lactating females.
6. Have a history of epilepsy or serious head injury.
7. Have a known history of long QT syndrome or cardiac tachy-arrhythmia.
8. Have hypersensitivity to any corticotropin releasing hormone antagonists.
9. Test positive at screening for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV), or have a history of a positive result.
10. Have a recent history (≤1 year) of alcohol or drug abuse, or current evidence of substance dependence or abuse criteria.
11. Used any anticoagulants or antiplatelet therapies within 30 days before screening.
12. Have an active bleeding disorder.
13. Used any other investigational drug within 30 days before initial screening, or plans to use an investigational drug (other than the study drug) during the study.
14. Have a blood loss ≥550 mL or donated blood within 56 days or donated plasma within 7 days before baseline.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (6):
- United States (6):
  - Neurocrine Clinical Site, Aurora, Colorado
  - Neurocrine Clinical Site, Indianapolis, Indiana
  - Neurocrine Clinical Site, Ann Arbor, Michigan
  - Neurocrine Clinical Site, Minneapolis, Minnesota
  - Neurocrine Clinical Site, Philadelphia, Pennsylvania
  - Neurocrine Clinical Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auchus RJ, Sarafoglou K, Fechner PY, Vogiatzi MG, Imel EA, Davis SM, Giri N, Sturgeon J, Roberts E, Chan JL, Farber RH. Crinecerfont Lowers Elevated Hormone Markers in Adults With 21-Hydroxylase Deficiency Congenital Adrenal Hyperplasia. J Clin Endocrinol Metab. 2022 Feb 17;107(3):801-812. doi: 10.1210/clinem/dgab749. PMID 34653252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study followed a sequential cohort design with four NBI-74788 dosing regimens, each administered for 14 consecutive days. There was ~2-week period to evaluate safety and tolerability data before proceeding from Cohort 1 to Cohort 2. Subjects who previously completed the study in Cohort 1 or 2 (and had no safety concerns) could reenroll into Cohorts 3 and/or 4 (in addition to new subjects); 18 unique subjects participated. First subject enrolled: 4/10/2018; Last subject completed: 4/7/2020
Period: Cohort 1 (50 mg QHS)
Arm/Group | Cohort 1 (50 mg QHS) | Cohort 2 (100 mg QHS) | Cohort 3 (100 mg QPM) | Cohort 4 (100 mg BID)
Started | 8 | 0 | 0 | 0
Completed | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2 (100 mg QHS)
Arm/Group | Cohort 1 (50 mg QHS) | Cohort 2 (100 mg QHS) | Cohort 3 (100 mg QPM) | Cohort 4 (100 mg BID)
Started | 0 | 7 | 0 | 0
Completed | 0 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 3 (100 mg QPM)
Arm/Group | Cohort 1 (50 mg QHS) | Cohort 2 (100 mg QHS) | Cohort 3 (100 mg QPM) | Cohort 4 (100 mg BID)
Started (Cohort 3 included 8 subjects who had participated in other cohorts.) | 0 | 0 | 8 | 0
Completed | 0 | 0 | 8 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 4 (100 mg BID)
Arm/Group | Cohort 1 (50 mg QHS) | Cohort 2 (100 mg QHS) | Cohort 3 (100 mg QPM) | Cohort 4 (100 mg BID)
Started (Cohort 4 included 5 subjects who had participated in other cohorts.) | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (50 mg QHS) | Cohort 2 (100 mg QHS) | Cohort 3 (100 mg QPM) | Cohort 4 (100 mg BID) | Total
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: A total of 18 unique subjects participated in the study. Subjects could participate in more than one cohort; Cohort 3 included 8 subjects and Cohort 4 included 5 subjects who had participated in other cohorts.
  years
    Cohort 1 (50 mg QHS): number analyzed (Participants) | 8 | 0 | 0 | 0 | 8
    Cohort 1 (50 mg QHS) | 31.1 (9.4) |  |  |  | 31.1 (9.4)
    Cohort 2 (100 mg QHS): number analyzed (Participants) | 0 | 7 | 0 | 0 | 7
    Cohort 2 (100 mg QHS) |  | 32.9 (9.7) |  |  | 32.9 (9.7)
    Cohort 3 (100 mg QPM): number analyzed (Participants) | 0 | 0 | 8 | 0 | 8
    Cohort 3 (100 mg QPM) |  |  | 30.9 (10.5) |  | 30.9 (10.5)
    Cohort 4 (100 mg BID): number analyzed (Participants) | 0 | 0 | 0 | 8 | 8
    Cohort 4 (100 mg BID) |  |  |  | 28.8 (8.2) | 28.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 18 unique subjects participated in the study. Subjects could participate in more than one cohort; Cohort 3 included 8 subjects and Cohort 4 included 5 subjects who had participated in other cohorts.
  Participants
    Cohort 1 (50 mg QHS): number analyzed (Participants) | 8 | 0 | 0 | 0 | 8
    Cohort 1 (50 mg QHS): Female | 4 |  |  |  | 4
    Cohort 1 (50 mg QHS): Male | 4 |  |  |  | 4
    Cohort 2 (100 mg QHS): number analyzed (Participants) | 0 | 7 | 0 | 0 | 7
    Cohort 2 (100 mg QHS): Female |  | 5 |  |  | 5
    Cohort 2 (100 mg QHS): Male |  | 2 |  |  | 2
    Cohort 3 (100 mg QPM): number analyzed (Participants) | 0 | 0 | 8 | 0 | 8
    Cohort 3 (100 mg QPM): Female |  |  | 3 |  | 3
    Cohort 3 (100 mg QPM): Male |  |  | 5 |  | 5
    Cohort 4 (100 mg BID): number analyzed (Participants) | 0 | 0 | 0 | 8 | 8
    Cohort 4 (100 mg BID): Female |  |  |  | 5 | 5
    Cohort 4 (100 mg BID): Male |  |  |  | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 18 unique subjects participated in the study. Subjects could participate in more than one cohort; Cohort 3 included 8 subjects and Cohort 4 included 5 subjects who had participated in other cohorts.
  Participants
    Cohort 1 (50 mg QHS): number analyzed (Participants) | 8 | 0 | 0 | 0 | 8
    Cohort 1 (50 mg QHS): Hispanic or Latino | 1 |  |  |  | 1
    Cohort 1 (50 mg QHS): Not Hispanic or Latino | 7 |  |  |  | 7
    Cohort 1 (50 mg QHS): Unknown or Not Reported | 0 |  |  |  | 0
    Cohort 2 (100 mg QHS): number analyzed (Participants) | 0 | 7 | 0 | 0 | 7
    Cohort 2 (100 mg QHS): Hispanic or Latino |  | 0 |  |  | 0
    Cohort 2 (100 mg QHS): Not Hispanic or Latino |  | 7 |  |  | 7
    Cohort 2 (100 mg QHS): Unknown or Not Reported |  | 0 |  |  | 0
    Cohort 3 (100 mg QPM): number analyzed (Participants) | 0 | 0 | 8 | 0 | 8
    Cohort 3 (100 mg QPM): Hispanic or Latino |  |  | 1 |  | 1
    Cohort 3 (100 mg QPM): Not Hispanic or Latino |  |  | 7 |  | 7
    Cohort 3 (100 mg QPM): Unknown or Not Reported |  |  | 0 |  | 0
    Cohort 4 (100 mg BID): number analyzed (Participants) | 0 | 0 | 0 | 8 | 8
    Cohort 4 (100 mg BID): Hispanic or Latino |  |  |  | 0 | 0
    Cohort 4 (100 mg BID): Not Hispanic or Latino |  |  |  | 8 | 8
    Cohort 4 (100 mg BID): Unknown or Not Reported |  |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 18 unique subjects participated in the study. Subjects could participate in more than one cohort; Cohort 3 included 8 subjects and Cohort 4 included 5 subjects who had participated in other cohorts.
  Participants
    Cohort 1 (50 mg QHS): number analyzed (Participants) | 8 | 0 | 0 | 0 | 8
    Cohort 1 (50 mg QHS): American Indian or Alaska Native | 0 |  |  |  | 0
    Cohort 1 (50 mg QHS): Asian | 1 |  |  |  | 1
    Cohort 1 (50 mg QHS): Native Hawaiian or Other Pacific Islander | 0 |  |  |  | 0
    Cohort 1 (50 mg QHS): Black or African American | 0 |  |  |  | 0
    Cohort 1 (50 mg QHS): White | 7 |  |  |  | 7
    Cohort 1 (50 mg QHS): More than one race | 0 | 0 |  |  | 0
    Cohort 1 (50 mg QHS): Unknown or Not Reported | 0 |  |  |  | 0
    Cohort 2 (100 mg QHS): number analyzed (Participants) | 0 | 7 | 0 | 0 | 7
    Cohort 2 (100 mg QHS): American Indian or Alaska Native |  | 0 |  |  | 0
    Cohort 2 (100 mg QHS): Asian |  | 0 |  |  | 0
    Cohort 2 (100 mg QHS): Native Hawaiian or Other Pacific Islander |  | 0 |  |  | 0
    Cohort 2 (100 mg QHS): Black or African American |  | 0 |  |  | 0
    Cohort 2 (100 mg QHS): White |  | 7 |  |  | 7
    Cohort 2 (100 mg QHS): More than one race |  | 0 |  |  | 0
    Cohort 2 (100 mg QHS): Unknown or Not Reported |  | 0 |  |  | 0
    Cohort 3 (100 mg QPM): number analyzed (Participants) | 0 | 0 | 8 | 0 | 8
    Cohort 3 (100 mg QPM): American Indian or Alaska Native |  |  | 0 |  | 0
    Cohort 3 (100 mg QPM): Asian |  |  | 1 |  | 1
    Cohort 3 (100 mg QPM): Native Hawaiian or Other Pacific Islander |  |  | 0 |  | 0
    Cohort 3 (100 mg QPM): Black or African American |  |  | 0 |  | 0
    Cohort 3 (100 mg QPM): White |  |  | 7 |  | 7
    Cohort 3 (100 mg QPM): More than one race |  |  | 0 |  | 0
    Cohort 3 (100 mg QPM): Unknown or Not Reported |  |  | 0 |  | 0
    Cohort 4 (100 mg BID): number analyzed (Participants) | 0 | 0 | 0 | 8 | 8
    Cohort 4 (100 mg BID): American Indian or Alaska Native |  |  |  | 0 | 0
    Cohort 4 (100 mg BID): Asian |  |  |  | 0 | 0
    Cohort 4 (100 mg BID): Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0
    Cohort 4 (100 mg BID): Black or African American |  |  |  | 0 | 0
    Cohort 4 (100 mg BID): White |  |  |  | 8 | 8
    Cohort 4 (100 mg BID): More than one race |  |  |  | 0 | 0
    Cohort 4 (100 mg BID): Unknown or Not Reported |  |  |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Day 14 in 17-hydroxyprogesterone (17-OHP) Morning Window Averages
Description: Percent changes in 17-OHP were assessed through the collection of samples from 0600 hours to 1000 hours both prior to study drug administration (i.e., at baseline) and after 14 days of study drug dosing. The 3 samples collected during this morning window at each visit were averaged and used to determine the percent change from baseline.
Time Frame: Baseline and Day 14
Population: Pharmacodynamic (PD) analysis set, which includes all enrolled participants who received at least one dose of study drug and have at least one PD parameter measurement at baseline and at least one PD parameter measurement at the Day 14 visit.
Measure: Median (Inter-Quartile Range); unit: Percent (%)
Arm/Group | Cohort 1 (50 mg QHS) | Cohort 2 (100 mg QHS) | Cohort 3 (100 mg QPM) | Cohort 4 (100 mg BID)
Number analyzed (Participants) | 8 | 7 | 8 | 8
Percent (%) | -60 [-85 to -32] | -58 [-93 to 8] | -53 [-86 to -43] | -64 [-86 to -51]

2. Secondary Outcome: Percent Change From Baseline to Day 14 in Androstenedione Morning Window Averages
Description: Percent changes in androstenedione were assessed through the collection of samples from 0600 hours to 1000 hours prior to study drug administration (baseline) and after 14 days of study drug dosing. The 3 samples collected at each visit during this morning window were averaged and used to determine the change and percent change from baseline.
Time Frame: Baseline and Day 14
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent (%)
Arm/Group | Cohort 1 (50 mg QHS) | Cohort 2 (100 mg QHS) | Cohort 3 (100 mg QPM) | Cohort 4 (100 mg BID)
Number analyzed (Participants) | 8 | 7 | 8 | 8
Percent (%) | -21 [-55 to -7] | -42 [-70 to -23] | -51 [-70 to 50] | -64 [-68 to -52]

3. Secondary Outcome: Percent Change From Baseline to Day 14 in Adrenocorticotropic Hormone (ACTH) Morning Window Averages
Description: Percent changes in ACTH were assessed through the collection of samples from 0600 hours to 1000 hours prior to study drug administration (baseline) and after 14 days of study drug dosing. The 3 samples collected at each visit during this morning window were averaged and used to determine the change and percent change from baseline.
Time Frame: Baseline and Day 14
Population: Pharmacodynamic analysis set, which includes all enrolled participants who received at least one dose of study drug and have at least one PD parameter measurement at baseline and at least one PD parameter measurement at the Day 14 visit.
Measure: Median (Inter-Quartile Range); unit: Percent (%)
Arm/Group | Cohort 1 (50 mg QHS) | Cohort 2 (100 mg QHS) | Cohort 3 (100 mg QPM) | Cohort 4 (100 mg BID)
Number analyzed (Participants) | 8 | 7 | 8 | 8
Percent (%) | -54 [-75 to -32] | -63 [-80 to -39] | -64 [-87 to -3] | -66 [-78 to -47]

ADVERSE EVENTS:
Time Frame: Up to 7 weeks
Arm/Group | Cohort 1 (50 mg QHS) | Cohort 2 (100 mg QHS) | Cohort 3 (100 mg QPM) | Cohort 4 (100 mg BID)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 5/7 | 5/8 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (50 mg QHS) (N=8) | Cohort 2 (100 mg QHS) (N=7) | Cohort 3 (100 mg QPM) (N=8) | Cohort 4 (100 mg BID) (N=8)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 — Single event of cholelithiasis, occurring 34 days after the last dose of study drug, assessed by the investigator as moderate in intensity and unlikely to be related to treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (50 mg QHS) (N=8) | Cohort 2 (100 mg QHS) (N=7) | Cohort 3 (100 mg QPM) (N=8) | Cohort 4 (100 mg BID) (N=8)
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovulation pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03525886/Prot_SAP_000.pdf